CLINICAL TRIAL: NCT01240811
Title: Impact of Intrauterine Contraception on the Immune Environment of the Female Genital Tract
Brief Title: Study of Immune Cell Changes in the Genital Tract 2 Months After Initiation of an IUD for Contraception
Acronym: CHIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharon Achilles (Other)
Responsible Party: Sponsor-Investigator, Sharon Achilles, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO09100199
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Genital Tract Mucosal Immunity; Genital Tract Microflora
Keywords: intrauterine device; IUD; levonorgestrel; copper; CD4; CCR5; microflora

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control-No IUD (No Intervention): Healthy volunteers not at risk of pregnancy and not using any hormonal contraception.
- Levonorgestrel IUS (Experimental): Healthy volunteers seeking contraception with IUD. Randomized to LNG IUS.
  Interventions: Drug: IUD placement; Drug: Levonorgestrel IUD
- Copper T380A IUD (Experimental): Healthy volunteers seeking contraception with IUD. Randomized to Copper T380A IUD.
  Interventions: Drug: IUD placement; Drug: Copper T380A IUD

INTERVENTIONS:
Drug: IUD placement — Volunteer subjects who are not at risk of pregnancy because they are either surgically sterilized or heterosexually abstinent will be enrolled into the control group (no intervention). All other volunteers will be seeking an IUD for contraception and will be randomized to LNG-IUD (Mirena) or Copper IUD (ParaGard).
  Arms: Copper T380A IUD; Levonorgestrel IUS
Drug: Levonorgestrel IUD
  Other Names: Mirena IUD
  Arms: Levonorgestrel IUS
Drug: Copper T380A IUD
  Other Names: ParaGard IUD
  Arms: Copper T380A IUD

SUMMARY:
This pilot study is being performed to investigate the influence that starting contraception with an IUD has on the local immune cell populations and features, with a particular focus on the cells and cell-surface features that are important in HIV transmission (CD4 cells and CCR5 cell receptors).

Based on results from large epidemiologic studies there seems to be a consistent finding of slightly increased HIV acquisition in women who use hormonal contraception. It is not clear if this is due to a biological phenomenon or if it relates to a difference in sexual behaviors/risks of women on hormonal contraceptives.

The study hypothesis is that CD4 cells and CCR5 HIV-tropic receptor density increases within the upper and lower genital tract of women 2 months after placement of progestin-containing intrauterine devices for contraception as compared with women not using hormonal contraception.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant, healthy females who are seeking an IUD for contraception
2. Age 18-40 years, inclusive at the time of enrollment
3. History of regular menstrual cycles defined as occurring every 21-35 days when not using hormones and with a variation of typical cycle length of no more than 5 days
4. Willing and able to sign the informed consent and to comply with the study protocol

Inclusion criteria for healthy control subjects:

1. Non-pregnant, healthy females
2. Age 18-40 years, inclusive at the time of enrollment
3. History of regular menstrual cycles defined as occurring every 21-35 days when not using hormones and with a variation of typical cycle length of no more than 5 days
4. Willing and able to sign the informed consent and to comply with the study protocol
5. Prior surgical sterilization or heterosexually abstinent

Exclusion Criteria:

1. Use of any hormonal or intrauterine contraceptive method within the past two months
2. Use of DMPA within the past 10 months
3. Any of the following within the past two months:

   * Pregnancy or breastfeeding
   * Surgery/biopsy of the vulva, vagina, or cervix
   * History of STI
   * New sexual partner
4. Evidence of vaginal/pelvic infection on screening

   * Abnormal wet mount (see description above)
   * Pelvic exam findings clinically consistent with infection
   * Positive screen for Gc, Ct, or HIV (will be excluded post randomization)
5. Active HSV/ulcerative disease in the genital tract or perineum
6. History of immunosuppression (diabetes, HIV, chronic steroid use)
7. Use of vaginal product (N9, microbicide, douche, antifungal, steroid, or hormone) within the past 30 days
8. Use of any systemic or vaginal steroid or antibiotic within the past 30 days
9. Vaginal or anal intercourse within 1 week of sample collection
10. Heterosexual vaginal intercourse since last menses without condom use
11. History of hysterectomy
12. History of malignancy in the uterus or cervix
13. Uterine anomaly (bicornuate uterus, uterine septum, or uterine didelphys)
14. Allergy to copper and/or intolerance to levonorgestrel

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Achilles, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the medical clinic and our database of prior research participants. Public advertisements included listing on our website, letters to the database mailing list, flyers placed on local college campuses, mailings to faculty, internet postings on Craig's list, and informational booths at on or off campus fairs.
Period: Overall Study
Arm/Group | Control-No IUD | Levonorgestrel IUS | Copper T380A IUD
Started | 8 | 17 | 17
Completed | 8 | 16 | 16
Not Completed | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control-No IUD | Levonorgestrel IUS | Copper T380A IUD | Total
Number analyzed (Participants) | 8 | 17 | 17 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 17 | 17 | 42
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6) | 26 (6) | 27 (4) | 26 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 17 | 42
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 17 | 17 | 42

OUTCOME MEASURES:

1. Primary Outcome: %CD4 Expressing CCR5 HIV Co-receptor in the Cervix and Endometrium
Description: Change in CCR5 expression on T-lymphocytes 2 months after insertion of IUD (either hormonal LNG-IUD or non-hormonal Cu-IUD) in cervix and endometrium as measured by flow cytomety
Time Frame: 2 months
Population: All 40 participants who completed the study were included in the analysis. There were no lost-to-follow up participants. One participant withdrew and one participant was excluded post-enrollment. Both of these participants were replaced to fill our goal enrollment of 40 participants in the study.
Measure: Mean (Standard Deviation); unit: % of T-cells expressing CCR5
Arm/Group | Control-No IUD | Levonorgestrel IUS | Copper T380A IUD
Number analyzed (Participants) | 8 | 16 | 16
% of T-cells expressing CCR5 | 4.9 (17.2) | 11.7 (29.8) | 7.2 (32.8)
Statistical Analysis 1: Comparison: Control-No IUD vs Levonorgestrel IUS; Test type: Superiority or Other; p = 0.80, ANOVA
Statistical Analysis 2: Comparison: Control-No IUD vs Copper T380A IUD; Test type: Superiority or Other; p = 0.97, ANOVA

2. Secondary Outcome: Change in Vaginal Flora
Description: Changes in vaginal flora as assessed by Nugent score The Nugent score is calculated by microscopically assessing for the presence of large Gram-positive rods (Lactobacillus morphotypes; decrease in Lactobacillus scored as 0 to 4), small Gram-variable rods (Gardnerella vaginalis morphotypes; scored as 0 to 4), and curved Gram-variable rods (Mobiluncus spp. morphotypes; scored as 0 to 2) and can range from 0 to 10. A score of 7 to 10 is consistent with bacterial vaginosis, 4-6 is consistent with intermediate vaginal flora, and 0-3 is normal vaginal flora.
Time Frame: 2 Months
Measure: Median (Full Range); unit: units on a scale
Groups:
- Levonorgestrel IUS: Healthy volunteers seeking contraception with IUD. Randomized to LNG IUS.
  IUD placement: Volunteer subjects who are not at risk of pregnancy because they are either surgically sterilized or heterosexually abstinent will be enrolled into the control group (no intervention). All other volunteers will be seeking an IUD for contraception and will be randomized to LNG-IUD (Mirena) or Copper IUD (ParaGard).
  Levonorgestrel IUD
- Copper T380A IUD: Healthy volunteers seeking contraception with IUD. Randomized to Copper T380A IUD.
  IUD placement: Volunteer subjects who are not at risk of pregnancy because they are either surgically sterilized or heterosexually abstinent will be enrolled into the control group (no intervention). All other volunteers will be seeking an IUD for contraception and will be randomized to LNG-IUD (Mirena) or Copper IUD (ParaGard).
  Copper T380A IUD
Arm/Group | Control-No IUD | Levonorgestrel IUS | Copper T380A IUD
Number analyzed (Participants) | 8 | 15 | 16
units on a scale | 0 [-7 to 2] | 1 [-3 to 6] | 0 [-8 to 5]
Statistical Analysis 1: Comparison: Control-No IUD vs Levonorgestrel IUS vs Copper T380A IUD; Difference in paired change in Nugent score from baseline to 2 months; Test type: Superiority; p = 0.08, Kruskal-Wallis

3. Secondary Outcome: Change in Quantities of Vaginal H2O2-producing Lactobacillus Species and Gardnerella Vaginalis
Description: Changes in vaginal flora as assessed by qPCR quantitation of H2O2 producing Lactobacilli species and Gardnerella vaginalis. Quantitative PCR (qPCR) results are reported as log concentration of gene copies/swab specimen.
Time Frame: 2 Months
Measure: Median (Full Range); unit: log gene copies/swab
Arm/Group | Control-No IUD | Levonorgestrel IUS | Copper T380A IUD
Number analyzed (Participants) | 8 | 15 | 16
log gene copies/swab
  Change in log Lactobacilli quantity | -0.6 [-4.5 to 3.1] | -0.1 [-8.3 to 1.0] | 0.1 [-3.1 to 5.1]
  Change in log Garnerella vaginalis quantity | 0 [-4.0 to 5.1] | 0 [-5.1 to 5.9] | 0 [-7.1 to 5.5]
Statistical Analysis 1: Comparison: Control-No IUD vs Levonorgestrel IUS vs Copper T380A IUD; Change in quantity of H2O2 producing Lactobacilli species by qPCR; Test type: Superiority; p = 0.46, Kruskal-Wallis
Statistical Analysis 2: Comparison: Control-No IUD vs Levonorgestrel IUS vs Copper T380A IUD; Change in quantity of Garnerella vaginalis species by qPCR; Test type: Superiority; p = 0.62, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | Control-No IUD | Levonorgestrel IUS | Copper T380A IUD
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/8 | 0/17 | 0/17

LIMITATIONS AND CAVEATS:
We identified a need for methods optimization prior to proceeding with a large definitive study to determine contraceptive hormone induced changes in genital tract immune cell populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No